CLINICAL TRIAL: NCT06324292
Title: Effect Of Digital Smile Design on Quality Of Life In Complete Denture Wearers: Randomized Clinical Trial
Brief Title: Effect Of Digital Smile Design on Quality Of Life In Complete Denture Wearers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Mostafa Abdelfatah, associate professor of oral and maxillofacial prosthodontics, Ain Shams University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: FDASU-RecID112324
Record Dates: First submitted 2024-03-15; First posted 2024-03-21 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Complete Edentulism
MeSH Terms: interventions — Denture, Complete

STUDY DESIGN:
Intervention Model Description: The participants allocated into two groups; a conventional denture followed by a digital group (CG) and a digital denture followed by a conventional one group (DG).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional denture followed by a digital one (Active Comparator): the participants will receive a conventional complete denture followed by a digital one having digital smile design
  Interventions: Procedure: complete denture, CG
- Digital denture followed by a conventional one (Active Comparator): the participants will receive a digital complete denture having digital smile design followed by a conventional one
  Interventions: Procedure: complete denture, DG

INTERVENTIONS:
Procedure: complete denture, CG — fabrication of conventional complete denture followed by a digital denture
  Arms: conventional denture followed by a digital one
Procedure: complete denture, DG — fabrication of digital complete denture followed by a conventional one
  Arms: Digital denture followed by a conventional one

SUMMARY:
The aim of the current study protocol is to compare the effect of two complete dentures made for completely edentulous patients; one digitally constructed using digital smile design (DSD) and another one conventionally constructed on the patient's quality of life and patient's satisfaction.

It is a clinical trial in which two dentures will be made for each patient, one will be digitally constructed using digital smile design (DSD) and the other one using the conventional method with a washout period of 3 weeks. Each patient will receive a questionnaire "Oral Health Impact Profile -19" (OHIP -19) for the edentulous patients to evaluate his satisfaction with the denture.

DETAILED DESCRIPTION:
Although the aesthetic results of digitally constructed dentures might be satisfactory for the patients, there is still little clinical evidence for the effect of using digital smile design DSD in denture construction on the patient's satisfaction. So, the objective of the current study is to find the effect of digital smile design (DSD) on quality of life in complete denture wearers compared to the conventionally created one. The current study is planned to be a crossover randomized Controlled Trial (RCT). The principal investigator, participants and the statistician will be blinded. Simple randomization of the patients in the will take place using a computer generated list (Software informer, Informer Technologies Inc) and allocated into two groups; a conventional denture followed by a digital group (CG) and a digital denture followed by a conventional one group (DG). Parallel allocation in ratio 1:1 will take place. The names of the participants in both groups will be placed in closed opaque sealed envelopes according to the computer generated list of random numbers and an envelope will be allocated to each patient. For blinding and allocation concealment, a third party rather than the authors and participants will be the only one to know the key so that the authors and the participants won't know in which group the participant will be. Afterwards, the authors will be informed by the randomization to be tabulated.

ELIGIBILITY:
Inclusion Criteria:

* completely edentulous patients
* well formed edentulous ridge
* healthy, pink, non edematous mucosa of even thickness

Exclusion Criteria:

* heavy smokers
* patients with parafunctional habits, temporomandibular joint disorders or orofacial motor disorders
* patients with physicological or psychiatric condition

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
quality of life assessment | 3 months
  OHIP-19 questionnaires for the edentulous patient will be used. A likert scale from 0 to 5 will be employed which zero will denote the ' very bad" experience with the denture and 5 will denote the "excellent" experience

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed MA Mohamed, BDS MSc MD, Study Chair — Ain Shams University
Locations (2):
- Egypt (2):
  - Faculty of Dentistry Ain Shams University, Cairo
  - Faculty of Dentistry, Ain Shams University, Cairo

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and statistical analysis plan will be available matching the criteria of the journal. However, data will be available from the corresponding author upon request once the paper is published.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study protocol and statistical analysis plan will be available matching the criteria of the journal. However, data will be available from the corresponding author upon request once the paper is published.
Access Criteria: data will be available from the corresponding author upon request once the paper is published.